CLINICAL TRIAL: NCT04115787
Title: Conservative Management in Patients Diagnosed With Grade 2 or Grade 3 CIN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CIN-2019-50
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: High-Grade Squamous Intraepithelial Lesions; Neoplasm Regression, Spontaneous; Disease Progression; Papillomavirus Infections
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Neoplasm Regression, Spontaneous; Disease Progression; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Consecutive inclusion and collection of information for all women attending the Cervical Disease Unit with an histological diagnosis of grade 2 or grade 3 CIN during the last 5 years, from January 2012 to December 2016, which meet the inclusion criteria, have voluntarily manifested pregnancy intendedness and had a minimum follow-up time of 2 years and a maximum of 7.

The aim is to evaluate whether the HSIL resolution rates (CIN 2 or CIN 3) are sufficient to support conservative management.

DETAILED DESCRIPTION:
Follow-up is performed every 4 months with colposcopy, cytology and biopsies. Colposcopy and cytology are performed for all control subjects. The need for biopsy is established according to the colposcopy exam findings to confirm H-SIL or cervical cancer. Follow-up is spaced every 6 months if the cytology and biopsy results indicate L-SIL / ASCUS in agreement with the colposcopic image. HPV tests are performed every 8-12 months. This strategy is maintained until the resolution of the H-SIL.

The conservative management stops if the H-SIL lesion persists after 24 months of follow-up, if the inclusion criteria are no longer met or if the exclusion ones are met.

Inclusion and exclusion criteria are reviewed at each visit and the conservative management ceases in case the patient decides to undergo conization.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age and willing to get pregnant in the future
* Acceptance of conservative management
* Commitment to study visits.
* Colposcopy with zone of transformation (ZT) type 1 or 2 (Unio esco-columnar totally visible) with image compatible with H-SIL and visible in its entirety.

Exclusion Criteria:

* Pregnant women
* Immunosuppression for human immunodeficiency virus (HIV) or iatrogenic type
* suspicion or diagnosis of Glandular Cell Atipia (ACG), Adenocarcinoma in situ (AIS) or cervical cancer (CC)
* Provided that inclusion criteria are not met

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women attending the Cervical Disease Unit with an histological diagnosis of grade 2 or grade 3 CIN during the last 5 years, from January 2012 to December 2016, which meet the inclusion criteria, have voluntarily manifested pregnancy intendedness and had a minimum follow-up time of 2 years and a maximum of 7.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2019-10-14 (Estimated); Primary Completion 2019-11-28 (Estimated); Study Completion 2019-12-28 (Estimated)

PRIMARY OUTCOMES:
H-SIL Resolution | 24 months
  In cases where H-SIL (cytologic, histological and colposcopic) is no longer detected during follow-up.
  Include the strict resolution, indulgent resolution and regression
H-SIL Regression | 24 months
  H-SIL is not detected, but with a low grade cytological, histologic or colposcopic lesion

SECONDARY OUTCOMES:
Factors probably related to the resolution | 24 months
  Demographics (age and origin), viral type, cytology, biopsy and colposcopy will be recorded at the beginning and end of the follow-up, as well as time until resolution, regression or progression and conization result.
Strict resolution | 24 months
  Negative HPV determination or different from the initial
Lenient resolution | 24 months
  Colposcopy lesion disappearance, negative results on cytology and biopsies with persistence of the same viral type of high initial grade.
Conization surgery | 24 months
  Patients undergoing surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Nerea Luqui Scarcelli, Barcelona, Spain